CLINICAL TRIAL: NCT03468959
Title: Maternal Polyunsaturated Fatty Acids in Association With Child Autism Spectrum Disorder in the MARBLES Study
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 225645
Record Dates: First submitted 2018-02-09; First posted 2018-03-19 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2018-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mother-child pairs: Families were recruited from lists of children receiving autism services obtained via the California Department of Developmental Services (DDS), from other studies at the Medical Investigation of Neurodevelopmental Disorders (MIND) Institute, or by self-referrals. The inclusion criteria were: a) mother or father had a biological child with ASD, and the mother was b) at least 18 years old; c) pregnant or planning a pregnancy, and biologically able to become pregnant; d) living within 2 hours of the MIND Institute; e) sufficiently fluent in English.
  Interventions: Behavioral: Maternal Supplemental PUFA Intake

INTERVENTIONS:
Behavioral: Maternal Supplemental PUFA Intake — Maternal Supplemental PUFA Intake included sources from the questionnaires and plasma

SUMMARY:
This study is to examine the association between maternal omega3 and other polyunsaturated fatty acids (PUFAs) during pregnancy and autism spectrum disorder (ASD) as well as other non-typical development (Non-TD) in the prospective Markers of Autism Risk in Babies-Learning Early Signs (MARBLES) cohort.

ELIGIBILITY:
Inclusion Criteria:

* Mother or father had a biological child with ASD
* Mother is at least 18 years old
* Mother is pregnant or planning a pregnancy, and biologically able to become pregnant
* Mother is living within 2 hours of the MIND Institute
* Mother is sufficiently fluent in English

Exclusion Criteria:

* Mothers with diseases which will influence on their study participation

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families were recruited from lists of children receiving autism services obtained via the California Department of Developmental Services (DDS), from other studies at the Medical Investigation of Neurodevelopmental Disorders (MIND) Institute, or by self-referrals.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
autism spectrum disorder group (ASD) | 36 months
  number of people with ASD

SECONDARY OUTCOMES:
A group of typically development (TD) people | 36 months
  number of typically developed people

OTHER OUTCOMES:
A group of non-typical development (Non-TD) people | 36 months
  number of people with non-typical development